CLINICAL TRIAL: NCT04327531
Title: Evaluation of Covid 19 Knowledge Anxiety and Expectation Levels of Turkish Physicians, Survey Study
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: turkishcovid19
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; Physician-Patient Relations
Keywords: covid-19; turkish physicians
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: turkish physicians — turkish physicians, who work active in pandemic hospital.

SUMMARY:
It is aimed to measure the general health information of Turkish physicians about covid 19 pandemic, to evaluate anxiety levels and to evaluate future expectations in this period.

ELIGIBILITY:
Inclusion Criteria:

* turkish physicians
* work active in pandemic hospital

Exclusion Criteria:

* work in another country
* retired physicians

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: turkish physicians, who work active in pandemic hospital
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of covid-19 knowledge level of turkish physicians | 1 month
  beck depression scale
  The BDI inventory has maximum of 63 and minimum of 0 scores:
  (0-10): Are considered normal ups and downs (11-16): Mild mood disturbance (17-20): Borderline clinical depression (21-30): Moderate depression, (31-40): Severe depression, Over 40: Extreme depression. A persistent score of !17, requires psychiatric treatment

SECONDARY OUTCOMES:
what they think about the future | 1 month
  Turkish physicians write their thoughts about the health system after covid 19 with their own sentences

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Yalcin Bahat P, Aldikactioglu Talmac M, Bestel A, Topbas Selcuki NF, Karadeniz O, Polat I. Evaluating the effects of the COVID-19 pandemic on the physical and mental well-being of obstetricians and gynecologists in Turkey. Int J Gynaecol Obstet. 2020 Oct;151(1):67-73. doi: 10.1002/ijgo.13287. Epub 2020 Aug 11. PMID 32602562